CLINICAL TRIAL: NCT00208767
Title: Effect of Valsartan on Endothelial Function, Oxidative Stress, Carotid Atherosclerosis, and Endothelial Progenitor Cells (EFFERVESCENT)
Brief Title: Effect of Valsartan on Carotid Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor of Medicine, Emory University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00024913; CVAL489AUS51 (Other: Other)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Carotid Artery Diseases; Atherosclerosis
Keywords: Angiotensin receptor blockade; Oxidative stress; Endothelial dysfunction
MeSH Terms: conditions — Carotid Artery Diseases; Atherosclerosis | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan (Active Comparator): Valsartan titrated up to 320 mg orally daily
  Interventions: Drug: Valsartan
- Placebo (Placebo Comparator): Patients received a placebo instead of Valsartan
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valsartan — Valsartan was titrated to a target dose of 320 mg orally daily
  Other Names: Diovan is a brand name of Valsartan
  Arms: Valsartan
Drug: Placebo — A matched placebo pill will be given orally daily.
  Arms: Placebo

SUMMARY:
The EFFERVESCENT trial is designed to evaluate the effects of a specific ARB, called valsartan, on atherosclerosis. The investigators want to know if treatment with valsartan will increase the blood levels of markers responsible for repair of the vessel wall, reduce oxidation and inflammation, improve the function of the blood vessels, and arrest or slow down the progression of atherosclerosis over time.

DETAILED DESCRIPTION:
Atherosclerosis or 'hardening of the arteries' is a process that ultimately leads to the development of heart attacks, strokes, poor circulation, and death. Millions of Americans are affected by this progressive disease of the arteries. Researchers have tried to understand the very complex processes that lead to hardening of the arteries. Part of this research has taught the investigators that there are specific molecules that can cause damage or injury to the vessel wall by increasing oxidation and inflammation which, in turn, leads to atherosclerosis. Other molecules and cells have been found that can actually repair the vessel wall.

Currently, the best treatment the investigators have for preventing or slowing atherosclerosis is to control the patients' risk factors such as high blood pressure, diabetes, or cholesterol levels using prevention and specific drugs. Angiotensin receptor blockers (ARBs) are a class of drugs that have been shown in clinical trials to have many beneficial effects in patients with high blood pressure, advanced heart diseases (such as after heart attack and heart failure), and diabetes. However, whether these drugs will also be useful in people with early signs of hardening of the arteries, measured as a thickening of the carotid (neck) arteries is unknown, and is the purpose of this study.

The EFFERVESCENT trial is designed to evaluate the effects of a specific ARB, called valsartan, on atherosclerosis. The investigators want to know if treatment with valsartan will increase the blood levels of markers responsible for repair of the vessel wall, reduce oxidation and inflammation, improve the function of the blood vessels, and arrest or slow down the progression of atherosclerosis over time.

In this study, the investigators will recruit subjects who have a hardening or thickening of their carotid arteries, one of the main blood vessels in the neck. People will be screened with ultrasound or sonar examination for this. Two-thirds of those eligible for participation will receive valsartan while the remaining one-third will receive a placebo pill. The investigators and subjects will be unaware of which drug is being given until the end of the study. The study will last for 2 years. Half of the individuals will also be treated with a statin drug (used for cholesterol reduction) and the remaining individuals will not be on a statin.

The investigators will measure carotid artery thickening with magnetic resonance imaging (MRI); forearm blood vessel function using ultrasound; and they will perform blood tests to measure oxidation and inflammation in the blood stream and circulation stem cells that are responsible for healing. These tests will be repeated at 3 months, 1 year and 2 years after starting treatment. The investigators will also collect blood for genotyping where the DNA will be stored for future analysis to study whether subjects' genotype alters their susceptibility to treatments. The investigators' hypothesis is that ARB treated individuals will have less oxidation and inflammation, higher levels of stem cells, and a slower progression of arterial thickening.

Finding an early treatment for atherosclerosis would hopefully prevent future strokes, heart attacks, and deaths leading to improved longevity and reduced medical expenditure.

ELIGIBILITY:
Inclusion Criteria:

* > 0.65 mm intima-media thickness of the carotid artery measured by ultrasound
* Males aged 21-80 years or women without child bearing potential up to age 80
* Can be on concomitant therapy with aspirin, thiazide diuretics, calcium antagonists (for treatment of hypertension), or beta-receptor antagonists.
* May be on statin if on stable dose for at least 2 months before recruitment

Exclusion Criteria:

* Angiotensin-converting enzyme (ACE) inhibitor or ARB therapy in the previous 3 months.
* Initiation or change in dose of statin therapy within 2 months before the study
* Inability to return to Emory for follow-up blood drawing and MR imaging
* Age < 21 or > 80 years
* Premenopausal females with potential for pregnancy
* Current neoplasm
* Chronic renal failure [creatinine > 2.5 mg/dL]
* Diabetes with hemoglobin (Hb) A1c > 8.5
* Anticipated change in lipid lowering therapy
* Inability to give informed consent
* MR exclusion criteria
* Blood pressure > 140 mmHg systolic and > 90 mmHg diastolic
* Low-density lipoprotein (LDL) cholesterol level >130 mg/dl
* Acute coronary syndrome within 2 months
* Acute cerebrovascular accident within 2 months

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Emory Healthcare sites or by advertisement between March 2005 and October 2008.
Pre-assignment Details: 60 of the enrolled subjects were already on long-term statin therapy and were stratified for statin use before randomization. Subjects on statin therapy were switched to simvastatin 40 mg daily unless they were already on high dose statin therapy and thus were placed on 80 mg daily of simvastatin for the duration of the study.
Period: Overall Study
Arm/Group | Valsartan | Placebo
Started | 80 | 40
Completed | 53 | 33
Not Completed | 27 | 7
Not completed — Adverse Event | 9 | 1
Not completed — Withdrawal by Subject | 14 | 3
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan | Placebo | Total
Number analyzed (Participants) | 80 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9) | 62 (9) | 60 (9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 40 | 120
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 21 | 59
  Male | 42 | 19 | 61
Region of Enrollment [Number; unit: participants]
  United States | 80 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Vessel Wall Area (VMA) of the Carotid Bulb From Baseline to 2 Years
Description: The PI will measure carotid artery thickening with magnetic resonance imaging.
Time Frame: Baseline, 2 years
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Valsartan | Placebo
Number analyzed (Participants) | 49 | 27
mm2 | -6.7 (2.4) | 3.4 (3.1)

ADVERSE EVENTS:
Arm/Group | Valsartan | Placebo
Serious Adverse Events (participants affected / at risk) | 3/80 | 0/40
Other Adverse Events (participants affected / at risk) | 0/80 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valsartan (N=80) | Placebo (N=40)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
Majory injury/accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No